CLINICAL TRIAL: NCT05217303
Title: A Single-arm, Multi-center Phase II Clinical Study to Evaluate the Efficacy and Safety of HL-085 in Advanced Melanoma Patients With NRAS Mutation
Brief Title: HL-085 in NRAS-mutated Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-101-II
Record Dates: First submitted 2022-01-07; First posted 2022-02-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
Keywords: HL-085; MEK inhibitor; NRAS mutation; advanced melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HL-085 (Experimental): 12 mg BID HL-085
  Interventions: Drug: HL-085

INTERVENTIONS:
Drug: HL-085 — HL-085 capsule administered orally twice daily (BID) in a 21-day treatment cycle

SUMMARY:
This was an open-label, single-arm, multi-center phase II clinical study, aimed at investigating the efficacy and safety of HL-085 capsule in the treatment of advanced melanoma patients with NRAS mutation.

DETAILED DESCRIPTION:
This was an open-label, single-arm, multi-center phase II clinical study, aimed at investigating the efficacy and safety of HL-085 capsule in the treatment of advanced melanoma patients with NRAS mutation. The primary objective was to evaluate the objective response rate (ORR) of oral HL-085 capsule in patients with advanced melanoma harboring NRAS mutation. The secondary objectives were to evaluate the progression-free survival (PFS), disease control rate (DCR), duration of remission (DOR), 1-year survival rate, overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 Years or older (male or female).
* Patients have histologically or cytologically confirmed Unresectable stage III or IV melanoma;
* Able to provide the genetic test report with documented NRAS mutation at baseline.
* At least one target lesion as per RECIST v1.1 criteria.
* Previous chemotherapy, immunotherapy, or radiotherapy must have been completed at least 4 weeks prior to study drug administration, and all related toxic reactions (with the exception of alopecia) must have been resolved (to Grade ≤1 or baseline) prior to study drug administration.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy > 3 months.
* No major surgery (excluding baseline tumor biopsy) or major trauma occurred at least 14 days prior to study drug administration.

Exclusion Criteria:

* Patients with active central nervous system (CNS) lesions (i.e., radiological evidence of instability, symptomatic lesions) should be excluded. Note: Patients receiving stereotactic brain radiotherapy or surgery who have shown no brain disease progression over a period of 3 months or longer are eligible for inclusion.
* Patients had received any other study treatment within the past 4 weeks prior to study drug administration.
* Inability to swallow the capsule, refractory nausea and vomiting, malabsorption, extracorporeal biliary shunt, or any small intestinal resection that would preclude adequate absorption of the study drug.
* ECG QTcB ≥ 480 msec (adjusted by Bazetts formula) during screening, or a history of congenital long QT syndrome.
* Bleeding symptoms of Grade 3 as defined by the National Cancer Institute General Terminology Standard for Adverse Events (NCI CTCAE V5.0) within the past 4 weeks prior to study initiation.
* One of the following situations occurs within the past 6 months prior to administration of study drug: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass grafting, symptomatic congestive heart failure, serious arrhythmia, uncontrolled hypertension, cerebrovascular accident, or transient ischemic attack, or symptomatic pulmonary embolism.
* Current use of other anti-cancer drugs (hormone therapy was acceptable).
* Uncontrolled concomitant diseases or infectious diseases.
* Patients have retinal vein occlusion (RVO), retinal pigment epithelial detachment (RPED) or other retinal diseases previously or currently.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-02-19 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | through study completion, an average of 1 year
  To evaluate the objective response rate (ORR) of patients with advanced melanoma harboring NRAS mutation. ORR by RECIST v1.1 following treatment with HL-085

SECONDARY OUTCOMES:
progression-free survival (PFS) | through study completion, an average of 1 year
  To evaluate the progression-free survival (PFS), disease control rate (DCR), duration of remission (DOR) of patients with advanced melanoma harboring NRAS mutation after HL-085 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, Ph.D, Study Director — Shanghai Kechow Pharma, Inc.
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Oncology Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No